CLINICAL TRIAL: NCT02051777
Title: Hospital Discharge Oral Nutrition Support Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NCC801
Record Dates: First submitted 2014-01-17; First posted 2014-01-31 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ONS 1 and DA (Other): Oral Nutritional Supplement 1 and Dietary Advice
  Interventions: Dietary Supplement: Oral Nutritional Supplement 1; Dietary Supplement: Dietary Advice
- ONS 2 and DA (Other): Oral Nutritional Supplement 2 and Dietary Advice
  Interventions: Dietary Supplement: Oral Nutritional Supplement 2; Dietary Supplement: Dietary Advice
- DA Alone (Other): Dietary Advice Alone
  Interventions: Dietary Supplement: Dietary Advice

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplement 1 — Containing macro and micronutrients
  Arms: ONS 1 and DA
Dietary Supplement: Oral Nutritional Supplement 2 — Containing macro and micronutrients
  Arms: ONS 2 and DA
Dietary Supplement: Dietary Advice

SUMMARY:
To investigate the effect of different strategies for managing malnutrition in the community

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 50 years and over
* Able to eat and drink without the need for altered texture fluids
* Identified at risk of disease related malnutrition
* Competent to provide written informed consent
* Willingness to take part in the study and to follow the study protocol

Exclusion Criteria:

* Individuals unable to eat or drink
* Chronic renal disease requiring dialysis
* Galactosaemia
* Dysphagia
* Normally or going to be residing in an institution e.g. care home upon discharge from hospital
* Palliative care
* Cancer (active treatment)
* Liver failure
* Poorly controlled diabetes
* Diagnosed lactose intolerance
* Participation in other clinical trials currently or in the previous 4 weeks
* Due to be discharged to an area out of the hospital region
* Requiring tube or parenteral nutrition
* Due to be discharged from hospital on oral nutrition support recommended by a Dietitian

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Nutrient Intake | 12 weeks (8 week intervention followed by 4 week follow up)
  Measured by 3 day diet diaries and 24 hour recall

CONTACTS AND LOCATIONS:
Locations (1):
- Nutricia Ltd, Bath, United Kingdom